CLINICAL TRIAL: NCT07311889
Title: Assessment of Patient Satisfaction and Healing Outcomes With the ELIXIR MD™ Device in the Perioperative Period of Plastic Surgery
Brief Title: Patient Satisfaction and Recovery Outcomes Associated With Perioperative ELIXIR MD Use
Status: Not yet recruiting | Type: Observational
Sponsor: Elixir MD Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ELIXIR-001
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain; Postoperative Edema; Postoperative Ecchymosis; Surgical Wound Healing; Postsurgical Recovery
Keywords: Photobiomodulation; Plastic Surgery; Postoperative Care; Patient-Reported Outcomes
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Perioperative photobiomodulation light therapy — Participants may receive perioperative light therapy as part of routine clinical care at the discretion of their treating clinician. The study does not assign, modify, or mandate the use of light therapy. Data are collected observationally to describe recovery outcomes associated with standard clinical practice.

SUMMARY:
The goal of this observational registry study is to characterize postoperative recovery outcomes in adult patients receiving standard-of-care perioperative light therapy using an FDA-cleared photobiomodulation device as part of routine clinical practice. The study aims to describe changes in patient-reported and clinician-assessed recovery measures following elective surgical procedures.

The main questions this registry aims to answer are:

1. How do patient-reported recovery outcomes, including pain, satisfaction, and perceived improvement, change over the postoperative period?
2. How do clinician-assessed indicators of recovery, such as swelling and bruising, change over time following surgery?

This study does not include a randomized comparison group. Outcomes will be described longitudinally within participants based on data collected during routine care.

Participants will:

1. Receive perioperative light therapy as part of standard clinical care, per their treating clinician
2. Complete patient-reported outcome questionnaires at defined postoperative time points
3. Undergo standardized clinical photography and routine clinical assessments as part of usual follow-up

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older undergoing elective plastic surgery (facial or body procedures) at a participating plastic surgery practice where the ELIXIR MD™ device is used as part of standard perioperative care.
* Able to provide informed consent and complete brief patient-reported questionnaires.

Exclusion Criteria:

* Pregnancy.
* Basal cell carcinoma, thyroid disorders, or malignant tumors.
* History of photosensitive skin disease or photosensitivity.
* Epilepsy or seizure disorders.
* Recent use of photosensitizing medications, including isotretinoin within the past 6 months; tetracyclines or ciprofloxacin within the past 5 days; chlorpromazine within the past 8 days; methotrexate within the past 3 days; or amiodarone, per physician discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years or older undergoing elective plastic surgery procedures (facial or body) at participating plastic surgery practices. All participants receive perioperative care in which the ELIXIR MD™ photobiomodulation device may be used as part of standard clinical practice, at the discretion of the treating surgeon. The registry enrolls patients across a range of procedure types and skin phototypes and collects de-identified patient-reported and clinical recovery data during routine perioperative follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported satisfaction with postoperative recovery | From baseline (preoperative) through 10 days postoperatively
  Patient-reported satisfaction with postoperative recovery assessed using a study-specific Global Satisfaction item adapted from Global Rating of Change (GROC) methodology. Responses are collected on a numeric Likert scale during routine postoperative follow-up and analyzed descriptively.
  Mean satisfaction score (0-10)
  % of patients reporting high satisfaction (≥7)

SECONDARY OUTCOMES:
Pain Intensity | From surgery through 10 days postoperatively
  Adapted from PROMIS Pain Intensity numeric rating scale
  PRS Description Pain intensity assessed using a numeric rating scale adapted from the PROMIS Pain Intensity measure (0-10). Scores are collected pre- and postoperatively and summarized descriptively as change from baseline.
  Unit Mean pain score Mean change from baseline
Global Rating of Change (Recovery) | From surgery through 10 days postoperatively
  Adapted from GROC (classic -5 to +5 format)
  Global recovery assessed using a Global Rating of Change (GROC) scale ranging from -5 (much worse) to +5 (very much better), capturing patient-perceived change in pain or healing compared to baseline.
  Unit Mean GROC score
  % reporting improvement (≥+2)
Swelling / Tightness / Bruising | Up to 10 days postoperatively
  Adapted from Common postoperative symptom severity NRS
  PRS Description Patient-reported swelling severity assessed using a study-specific numeric rating scale adapted from commonly used postoperative symptom severity measures.
  Unit Mean swelling score (1-5) Change from baseline
Scar Appearance & Symptoms | Up to 10 days postoperatively
  Adapted from Patient Scar Assessment Questionnaire (PSAQ - short form)
  Scar appearance and symptoms assessed using items adapted from the Patient Scar Assessment Questionnaire (PSAQ), including appearance, symptoms, awareness, and satisfaction domains.
  Unit Mean domain scores (1-5)
Return to Normal Activities | Up to 10 days postoperatively
  Adapted from Standard postoperative time-to-event self-report
  Time to return to usual daily activities assessed by patient-reported number of days from surgery to perceived return to baseline activity.
  Unit Days

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) generated in this observational registry, including patient-reported outcomes, procedure characteristics, and perioperative recovery assessments collected during routine clinical care. No direct identifiers will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning after publication of the primary study results and available upon reasonable request, with no predefined end date.
Access Criteria: Access to de-identified individual participant data (IPD) and supporting study documents will be limited to qualified researchers with a legitimate scientific purpose. Researchers may request access by submitting a written proposal to the sponsor describing the research question, analysis plan, and intended use of the data.
  Requests will be reviewed by the sponsor for scientific merit, feasibility, and compliance with ethical and privacy requirements. Approved researchers will be granted access only to de-identified participant-level data relevant to the approved proposal. No protected health information (PHI) will be shared.
  Data access will be provided through secure data transfer or controlled access methods, subject to execution of a data use agreement.

REFERENCES:
- [Background] Dompe C, Moncrieff L, Matys J, Grzech-Lesniak K, Kocherova I, Bryja A, Bruska M, Dominiak M, Mozdziak P, Skiba THI, Shibli JA, Angelova Volponi A, Kempisty B, Dyszkiewicz-Konwinska M. Photobiomodulation-Underlying Mechanism and Clinical Applications. J Clin Med. 2020 Jun 3;9(6):1724. doi: 10.3390/jcm9061724. PMID 32503238
- [Background] Jagdeo J, Austin E, Mamalis A, Wong C, Ho D, Siegel DM. Light-emitting diodes in dermatology: A systematic review of randomized controlled trials. Lasers Surg Med. 2018 Jan 22;50(6):613-28. doi: 10.1002/lsm.22791. Online ahead of print. PMID 29356026
- [Background] Karimi S, Sadeghi M, Amali A, Saedi B. Effect of Photobiomodulation on Ecchymosis after Rhinoplasty: A Randomized Single-Blind Controlled Trial. Aesthetic Plast Surg. 2020 Oct;44(5):1685-1691. doi: 10.1007/s00266-020-01760-9. Epub 2020 May 14. PMID 32410200
- [Background] Topaloglu N, Ozdemir M, Cevik ZBY. Comparative analysis of the light parameters of red and near-infrared diode lasers to induce photobiomodulation on fibroblasts and keratinocytes: An in vitro study. Photodermatol Photoimmunol Photomed. 2021 May;37(3):253-262. doi: 10.1111/phpp.12645. Epub 2020 Dec 23. PMID 33332651
- [Background] Serrage H , Heiskanen V , Palin WM , Cooper PR , Milward MR , Hadis M , Hamblin MR . Under the spotlight: mechanisms of photobiomodulation concentrating on blue and green light. Photochem Photobiol Sci. 2019 Aug 1;18(8):1877-1909. doi: 10.1039/c9pp00089e. Epub 2019 Jun 11. PMID 31183484
- [Background] Yadav A, Gupta A. Noninvasive red and near-infrared wavelength-induced photobiomodulation: promoting impaired cutaneous wound healing. Photodermatol Photoimmunol Photomed. 2017 Jan;33(1):4-13. doi: 10.1111/phpp.12282. PMID 27943458
- [Background] Baek WY, Byun IH, Yun IS, Kim JY, Roh TS, Lew DH, Kim YS. The effect of light-emitting diode (590/830 nm)-based low-level laser therapy on posttraumatic edema of facial bone fracture patients. J Craniomaxillofac Surg. 2017 Nov;45(11):1875-1877. doi: 10.1016/j.jcms.2017.08.027. Epub 2017 Sep 2. PMID 28986000
- [Background] Prado TP, Zanchetta FC, Barbieri B, Aparecido C, Melo Lima MH, Araujo EP. Photobiomodulation with Blue Light on Wound Healing: A Scoping Review. Life (Basel). 2023 Feb 18;13(2):575. doi: 10.3390/life13020575. PMID 36836932
- [Background] Hernandez-Bule ML, Naharro-Rodriguez J, Bacci S, Fernandez-Guarino M. Unlocking the Power of Light on the Skin: A Comprehensive Review on Photobiomodulation. Int J Mol Sci. 2024 Apr 19;25(8):4483. doi: 10.3390/ijms25084483. PMID 38674067
- [Background] Kuffler DP. Photobiomodulation in promoting wound healing: a review. Regen Med. 2016 Jan;11(1):107-22. doi: 10.2217/rme.15.82. Epub 2015 Dec 18. PMID 26681143